CLINICAL TRIAL: NCT05647317
Title: Design of a Mobile Technology-Based System for Patient Engagement and Physician-Directed Remote Management of Heart Failure
Brief Title: Mobile Technology-Based System for Patient Engagement and Physician-Directed Remote Management of Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alexander Sandhu, Instructor, CVMed, Department of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 67924
Record Dates: First submitted 2022-11-01; First posted 2022-12-12 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Heart Failure
Keywords: Heart Failure; Digital Health; Remote monitoring; Mobile Application
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital technology-based system for heart failure management (Other): This is a single-arm study to assess the feasibility and preliminary effectiveness of a digital technology-based system for heart failure management
  Interventions: Other: A combination of a provider-facing desktop and mobile application with a patient-facing mobile application

INTERVENTIONS:
Other: A combination of a provider-facing desktop and mobile application with a patient-facing mobile application — A combination of a provider-facing desktop and mobile application with a patient-facing mobile application that is integrated with a remote blood pressure cuff, heart rate monitor, and scale.

SUMMARY:
This pilot study is to assess the feasibility, preliminary utility and acceptance of a digital technology-based system for heart failure management.

DETAILED DESCRIPTION:
Heart failure continues to be a major public health problem. High-value, guideline-directed medical therapies (GDMT) for heart failure can reduce mortality and improve quality of life. However, large gaps in treatment with GDMT persist. While prior quality improvement efforts have focused on heart failure hospitalizations, there is a critical need to improve the quality-of-care post-discharge when the initiation and up-titration of GDMT is critical to optimizing outcomes. The main purpose of this pilot study is to assess the feasibility, preliminary utility and acceptance of a digital technology-based system for heart failure management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Diagnosis of heart failure
* Most recent left ventricular ejection fraction ≤ 40% in the prior year based on echocardiogram, MRI, CT, or nuclear perfusion
* Primary cardiologist enrolled in the study
* Currently admitted with upcoming discharge or discharged from hospital within the prior 2 weeks
* At least two eligible heart failure therapies (guideline-recommended BB, RASI, MRA, or SGLT2i) not yet initiated or on ≤ 50% of target dose

Exclusion Criteria:

* Receives dialysis
* Inotropic therapy during hospitalization
* History of heart transplant or actively listed on heart transplant waiting list
* History of left ventricular assist device implantation
* Cardiac amyloidosis
* Pregnant or currently trying to be pregnant
* Life expectancy estimated less than 6 months related to non-cardiac comorbidities as per investigator's judgement
* Actively enrolled in hospice or comfort care
* Currently participating in an investigational device or drug study or having participated in such a study within 30 days prior to screening
* Subject or their caregiver without a smartphone
* Subject or their caregiver not proficient with written and spoken English
* Subject unavailable to complete all study procedures (e.g., interviews) to the best of the subject and investigator's knowledge
* Any other disorder or condition that, in the opinion of the investigator would pose a risk to subject safety or interfere with the study evaluation, procedures or completion
* Subject has diminished decision-making capacity
* Planned discharge to skilled nursing facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-28 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Patient Acceptability of the intervention | At Study completion (12-week follow-up visit)
  The proportion of patients who assess the DOT-HF intervention as an acceptable method of post-discharge heart failure management. This will be assessed during a semi-structured interview between individual participants and a trained interviewer.
Patients' Engagement score | At Study completion (12-week follow-up visit)
  A weighted proportion of requested actions completed by the patient. These actions include daily blood pressure measurements, daily weight assessment, daily health status assessment, biweekly KCCQ-12 assessment, and review of educational videos and health summary data. The minimum score is 0% and maximum score is 100%.
Clinicians' Response to Notification | At Study completion (12-week follow-up visit)
  The proportion of DOT-HF clinician notifications that lead to a clinician response over the 12-week follow-up period. Each of the clinician DOT-HF notifications are detailed below. These include notification of eligible therapy adjustment, worsening patient-reported health status, and weight gain. Eligible clinician actions include medication changes or new telephone, video, or in-person clinic encounters in response to the notification.

SECONDARY OUTCOMES:
Proportion of days with weight assessed | At Study Completion (12-week follow-up visit)
  The proportion of days weight is recorded by the participant using the ENGAGE-HF app. The minimum is 0% and maximum is 100%.
Proportion of days with daily health status completed | At Study Completion (12-week follow-up visit)
  The proportion of days daily health status is recorded by the participant using the ENGAGE-HF app. The minimum is 0% and maximum is 100%.
Proportion of Kansas City Cardiomyopathy Questionnaire-12 assessments completed | At Study Completion (12-week follow-up visit)
  The proportion of biweekly periods that the Kansas City Cardiomyopathy Questionnaire-12 health status is recorded by the participant using the ENGAGE-HF app. The minimum is 0% and maximum is 100%.
Proportion of days with blood pressure (systolic) assessed | At Study Completion (12-week follow-up visit)
  The proportion of days blood pressure (systolic) is recorded by the participant using the ENGAGE-HF app. The minimum is 0% and maximum is 100%.
Proportion of days with medication adherence assessed | At Study Completion (12-week follow-up visit)
  The proportion of days medication adherence is recorded by the participant using the ENGAGE-HF app. The minimum is 0% and maximum is 100%.
Sustainability of DOT-HF technology for Patients | At 6 week, At Study Completion (12-week follow-up visit)
  Sustainability will also be assessed via semi-structured interview questions to assess patient's and clinician's interest in continuing to use the DOT-HF intervention.
Feasibility of DOT-HF technology for Patients | At Study Completion (12 week follow up visit)
  Feasibility will be assessed via semi-structured interview questions to assess barriers to use the DOT-HF intervention.
Utility of DOT-HF technology for Clinicians | At study completion (12 week follow up visit)
  Clinician perception of the utility of DOT-HF will be assessed based on clinician actions in response to DOT-HF notifications. We will assess each of the types of notifications aggregated in co-primary endpoint #3:
  * Notification of eligible therapy adjustment
  * Worsening patient-reported health status
  * Weight gain
  For each endpoint, we will separately evaluate the proportion of notifications that were followed by a medication adjustment and the proportion that were followed by a previously unplanned encounter between the clinician/clinic nurse and the patient.
Acceptability of DOT-HF technology for Clinicians | At study completion (12 week follow up visit)
  Clinician perception of the acceptability of DOT-HF will be assessed by clinician responses to a survey administered at the end of the study and semi-structured interview.
Generalizability of the DOT-HF Intervention | At study completion (12 week follow up visit)
  The generalizability of our study will be evaluated by comparing sociodemographic data between participants and eligible individuals who decline participation. Sociodemographics include age, gender, and race.
Guideline-Directed Medical Therapy Score | Baseline, At study completion (12 week follow-up visit)
  A score based on the heart failure medications prescribed. The minimum score is 0% and maximum score is 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Sandhu, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital & Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No